CLINICAL TRIAL: NCT06157060
Title: Prediction of Hepatocellular Carcinoma Recurrence After Curative Treatment by Longitudinal Monitoring Minimal Residual Disease Based on Circulating Tumor DNA
Brief Title: Prediction of Hepatocellular Carcinoma Recurrence After Curative Treatment by Longitudinal Monitoring MRD Based on ctDNA
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KY-232-01
Record Dates: First submitted 2023-11-23; First posted 2023-12-05 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma Resectable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with hepatocellular carcinoma: Patient with hepatocellular carcinoma who can undergo radical resection
  Interventions: Diagnostic Test: circulating tumor DNA

INTERVENTIONS:
Diagnostic Test: circulating tumor DNA — blood sample and tissue specimen for circulating tumor DNA will be done to patient with hepatocellular carcinoma

SUMMARY:
This study will conduct a prospective cohort study to verify the predictive value of ctDNA-MRD longitudinal monitoring model in predicting postoperative recurrence, verify whether ctDNA-MRD longitudinal monitoring model can indicate recurrence earlier than imaging examination, and explore the feasibility of guiding adjuvant therapy after curative treatment based on this model.

DETAILED DESCRIPTION:
The recurrence rate of hepatocellular carcinoma after curative treatment is high, and the minimal residual disease(MRD) in patients is the major cause of liver cancer recurrence, and the MRD is an important basis for the decision of adjuvant therapy after curative treatment. Previous studies have confirmed that circulating tumor DNA(ctDNA)-MRD monitoring model can accurately predict the recurrence of hepatocellular carcinoma patients. It was also found in retrospective analysis that tumor free survival was significantly prolonged after ctDNA-positive treatment for hepatocellular carcinoma after resection. This study will conduct a prospective cohort study to verify the predictive value of ctDNA-MRD longitudinal monitoring model in predicting postoperative recurrence, verify whether ctDNA-MRD longitudinal monitoring model can indicate recurrence earlier than imaging examination, and explore the feasibility of guiding adjuvant therapy after curative treatment based on this model.This study is to verify the predictive value of ctDNA-MRD longitudinal monitoring model in predicting postoperative recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-75 years;
2. Preoperative imaging examination diagnosed hepatocellular carcinoma (BCLC) stage 0 / stage A/stage B, eligible for radical surgery;
3. ECOG physical status score is 0-1;
4. Child-Pugh score is 5-6 points (Level A);
5. Not received any anti-tumor therapy;
6. Laboratory tests were at normal levels within 7 days before enrollment.

Exclusion Criteria:

1. Patient can't provide blood samples for ctDNA testing;
2. Patient with two or more types of tumors at the same time;
3. Non-primary liver lesions;
4. Pregnant or lactating women;
5. Patient with a history of other malignant tumors within the past 5 years or at the same time, except cured skin basal cell carcinoma, cervical carcinoma in situ and thyroid papillary carcinoma;
6. Patient with serious heart disease;
7. Other conditions deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hepatocellular carcinoma who can undergo radical surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | 2 years
  percentage of recurrence-free survival 2 years after surgery

SECONDARY OUTCOMES:
Correlation between ctDNA-MRD status dynamic changes and relapse | 2 years
  Correlation between ctDNA-MRD status dynamic changes and relapse

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Principal Investigator — Southern Medical University
Locations (7):
- China (7):
  - The Sixth Affiliated Hospital of South China University of Technology, Foshan, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Shunde Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong